CLINICAL TRIAL: NCT01549834
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of ABT-126 in Subjects With Mild to Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors
Brief Title: Evaluate the Efficacy and Safety of ABT-126 in Subjects With Mild to Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M11-793; 2011-004849-40 (EudraCT Number)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ABT-126

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ABT-126 Low Dose (Experimental): low dose
  Interventions: Drug: ABT-126
- ABT-126 High Dose (Experimental): high dose
  Interventions: Drug: ABT-126
- sugar pill (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ABT-126 — Low Dose
  Arms: ABT-126 Low Dose
Drug: ABT-126 — High Dose
  Arms: ABT-126 High Dose
Drug: placebo — Placebo
  Arms: sugar pill

SUMMARY:
This is an efficacy and safety study evaluating a new treatment for subjects with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
This is a Phase 2 study designed to evaluate the efficacy and safety of ABT-126 in approximately 420 adults with mild to moderate Alzheimer's disease who are taking stable doses of acetylcholinesterase inhibitors. Subjects will be randomized to one of two ABT-126 dose arms or placebo for a 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* The subject and caregiver must voluntarily sign and date an informed consent. If the subject does not have the capacity to provide informed consent, full informed consent must be obtained from the subject's representative and assent must be obtained from the subject.
* The subject is a male or female between the ages of 55 and 90 years, inclusive, at Screening Visit 1. Main Inclusion (Continued):
* The subject meets the Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable AD.
* The subject must be receiving a stable dose of an AChEI (donepezil or rivastigmine) for at least 90 days prior to Screening Visit 1.
* The subject has a Mini-Mental Status Examination (MMSE) total score of 12 to 24, inclusive, at Screening Visit 1.
* The subject has a Cornell Scale for Depression in Dementia (CSDD) score ≤ 10 at Screening Visit 1.
* The subject has a Modified Hachinski Ischemic Scale (MHIS) score of ≤ 4 at Screening Visit 1.
* With the exception of a diagnosis of mild-to-moderate Alzheimer's disease and the presence of stable medical conditions, the subject is in general good health, based upon the results of medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG).
* The subject has an identified, reliable caregiver who will provide support and ensure compliance with the study medication and procedures, and provide accurate information about the subject's status during the study.

Exclusion Criteria:

* The subject has taken galantamine or memantine within 60 days prior to Screening Visit 1.
* The subject has received excluded concomitant medications.
* The subject has clinically significant abnormal laboratory values at Screening Visit 1 as determined by the investigator.
* The subject has a history of any significant neurologic disease other than Alzheimer's disease including Parkinson's disease, multi-infarct or vascular dementia, Huntington's disease, normal pressure hydrocephalus, progressive supranuclear palsy, multiple sclerosis, any seizures, mental retardation or a history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
* In the opinion of the investigator, the subject has any clinically significant uncontrolled medical or psychiatric illness.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - cognitive subscale | Measurements up through 24 weeks
  An assessment tool which focuses on cognitive function and memory

SECONDARY OUTCOMES:
Mini Mental Status Exam | Measurements up through 24 weeks
  Questionnaire which provides a quantitative measure of cognition
Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) | Measurements up through 24 weeks
  Caregiver-based assessment of activities of daily living
DEMentia Quality of Life (DEMQOL) | Measurements up through 24 weeks
  Health-related quality of life measurement tool
Clinician Interview-Based Impression of Change - plus (CIBIC-plus) | Measurements up through 24 weeks
  Measures a global impression of change in severity of dementia
Neuropsychiatry Inventory (NPI) | Measurements up through 24 weeks
  Assesses the presence of psychopathology in subjects with Alzheimer's disease and other dementias
Partner-Patient Questionnaire for Shared Activities (PPQSA) | Measurements up through 24 weeks
  Measures the extent to which mood and mental state interferes with the patient-partner relationship
Resource Use in Dementia (RUD-Lite) | Measurements up through 24 weeks
  Brief measurement tool for resource utilization
EuroQol-5D Questionnaires | Measurements up through 24 weeks
  Assesses patient's mobility, self-care, usual activity, pain/discomfort and anxiety/depression
Wechsler Memory Scale-III (WMS-III) Working Memory Index | Measurements up through 18 weeks
  Assesses working memory

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gault, MD, Study Director — AbbVie
Locations (43):
- United States (11):
  - Site Reference ID/Investigator# 66528, Fresno, California
  - Site Reference ID/Investigator# 69602, Long Beach, California
  - Site Reference ID/Investigator# 66527, San Francisco, California
  - Site Reference ID/Investigator# 66530, Hamden, Connecticut
  - Site Reference ID/Investigator# 66522, Delray Beach, Florida
  - Site Reference ID/Investigator# 66524, Orlando, Florida
  - Site Reference ID/Investigator# 66531, Tampa, Florida
  - Site Reference ID/Investigator# 66529, West Palm Beach, Florida
  - Site Reference ID/Investigator# 66526, Elk Grove Village, Illinois
  - Site Reference ID/Investigator# 66525, Staten Island, New York
  - Site Reference ID/Investigator# 66523, Bennington, Vermont
- Canada (5):
  - Site Reference ID/Investigator# 71793, Gatineau
  - Site Reference ID/Investigator# 71794, Montreal
  - Site Reference ID/Investigator# 71798, Peterborough
  - Site Reference ID/Investigator# 71795, Toronto
  - Site Reference ID/Investigator# 71796, Verdun
- France (5):
  - Site Reference ID/Investigator# 71573, Dijon
  - Site Reference ID/Investigator# 77833, Limoges
  - Site Reference ID/Investigator# 68706, Paris
  - Site Reference ID/Investigator# 68704, Paris
  - Site Reference ID/Investigator# 68705, Toulouse
- Germany (6):
  - Site Reference ID/Investigator# 68768, Berlin
  - Site Reference ID/Investigator# 68764, Freiburg im Breisgau
  - Site Reference ID/Investigator# 68767, Hüttenberg
  - Site Reference ID/Investigator# 69960, Mittweida
  - Site Reference ID/Investigator# 68765, Munich
  - Site Reference ID/Investigator# 69959, Schwerin
- Greece (6):
  - Site Reference ID/Investigator# 68730, Athens
  - Site Reference ID/Investigator# 68732, Athens
  - Site Reference ID/Investigator# 68733, Athens
  - Site Reference ID/Investigator# 68731, Haidari, Athens
  - Site Reference ID/Investigator# 68729, Thessaloniki
  - Site Reference ID/Investigator# 68735, Thessaloniki
- South Africa (5):
  - Site Reference ID/Investigator# 67586, Belville
  - Site Reference ID/Investigator# 67582, Cape Town
  - Site Reference ID/Investigator# 67584, George
  - Site Reference ID/Investigator# 67585, Johannesburg
  - Site Reference ID/Investigator# 67583, Rosebank
- United Kingdom (5):
  - Site Reference ID/Investigator# 67787, Bath
  - Site Reference ID/Investigator# 67784, Glasgow
  - Site Reference ID/Investigator# 67786, London
  - Site Reference ID/Investigator# 67785, Manchester
  - Site Reference ID/Investigator# 67783, Warrington

REFERENCES:
- [Derived] Florian H, Meier A, Gauthier S, Lipschitz S, Lin Y, Tang Q, Othman AA, Robieson WZ, Gault LM. Efficacy and Safety of ABT-126 in Subjects with Mild-to-Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors: A Randomized, Double-Blind, Placebo-Controlled Study. J Alzheimers Dis. 2016;51(4):1237-47. doi: 10.3233/JAD-150978. PMID 26967214